CLINICAL TRIAL: NCT01351870
Title: A Prospective Randomised Controlled Trial of Hyperfractionated Versus Conventionally Fractionated Radiotherapy in Standard Risk Medulloblastoma
Brief Title: Hyperfractionated Versus Conventionally Fractionated Radiotherapy in Standard Risk Medulloblastoma (PNET4)
Acronym: SIOP-PNET-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC2003-06
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Medulloblastoma
MeSH Terms: conditions — Medulloblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Fractionation Regimen (Active Comparator): 1.8 Gy daily, 5 fractions per week
  Cranio-spinal axis:
  23.4 Gy in 13 fractions of 1.8 Gy
  Posterior fossa:
  30.6 Gy in 17 fractions of 1.8 Gy
  Interventions: Radiation: Standard Fractionation Regimen
- Hyperfractionated radiotherapy (Experimental): 1 Gy b.d. (minimum interval between fractions 8 hours). 10 fractions per week
  Craniospinal axis:
  36 Gy in 36 fractions of 1 Gy
  Posterior fossa:
  24 Gy in 24 fractions of 1 Gy
  Tumour Bed:
  8 Gy in 8 fractions of 1 Gy
  Interventions: Radiation: Hyperfractionated Radiotherapy

INTERVENTIONS:
Radiation: Standard Fractionation Regimen — 1.8 Gy daily, 5 fractions per week
  Cranio-spinal axis:
  23.4 Gy in 13 fractions of 1.8 Gy
  Posterior fossa:
  30.6 Gy in 17 fractions of 1.8 Gy
  Arms: Standard Fractionation Regimen
Radiation: Hyperfractionated Radiotherapy — 1 Gy b.d. (minimum interval between fractions 8 hours). 10 fractions per week
  Craniospinal axis:
  36 Gy in 36 fractions of 1 Gy
  Posterior fossa:
  24 Gy in 24 fractions of 1 Gy
  Tumour Bed:
  8 Gy in 8 fractions of 1 Gy
  Arms: Hyperfractionated radiotherapy

SUMMARY:
This is an international prospective randomised trial, which will compare two radiotherapy regimens in children and adolescents (aged 4 or 5 years to 21 years inclusive) with carefully staged 'standard risk' medulloblastoma.

DETAILED DESCRIPTION:
Patients eligible for the study will be those with non-metastatic medulloblastoma (by imaging and CSF cytology) at diagnosis. Patients randomised to the standard arm will receive conventionally fractionated (once a day) radiotherapy with a dose of 54 Gy to the posterior fossa and 23.4 Gy to the craniospinal axis. The experimental arm will be hyperfractionated (twice a day) radiotherapy (1 Gy b.d.) with a dose of 60 Gy to the posterior fossa with an additional 8 Gy to the tumour bed and 36 Gy to the craniospinal axis. Both groups will receive identical chemotherapy consisting of eight weekly doses of Vincristine given with radiotherapy and 8 courses of CCNU, cisplatin and vincristine following radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age at diagnosis at least 4 years or 5 years (according to the policy of the National Brain Tumour Group) and less than 22 years.
* Histologically proven medulloblastoma, including the following variants(WHO classification - 2000): classic medulloblastoma, nodular / desmoplastic medulloblastoma, melanotic medulloblastoma, medullomyoblastoma No CNS metastasis on MRI - supratentorial, arachnoid of the posterior fossa or spine.
* No clinical evidence of extra-CNS metastasis
* No tumour cells on the cytospin of lumbar CSF. Central Review of CSF cytology is recommended but not mandatory. It will be left to national policy.
* Radiotherapy to start no more than 40 days after surgery.
* Ability to receive twice daily radiotherapy.
* Vital functions within normal range for their age group.
* CTC grades < 2 for liver, renal, haematological and audiological function.
* No medical contraindication to radiotherapy or chemotherapy.
* Written informed consent (and patient assent where appropriate) according to the laws of each participating country. Written informed consent should also be sought for biological studies.
* National and local ethical committee approval according to the laws of each participating country (to include approval for biological studies).

Exclusion Criteria:

* One of the inclusion criteria is lacking.
* Brainstem or supratentorial primitive neuroectodermal tumour.
* Atypical teratoid rhabdoid tumour.
* Medulloepithelioma.
* Ependymoblastoma.
* Large cell médulloblastoma.
* Metastatic medulloblastoma (on CNS MRI and/or positive cytospin of postoperative lumbar CSF).
* Patient previously treated for a brain tumour or any type of malignant disease.
* Patients who are pregnant.
* Females who are sexually active and not taking reliable contraception.
* Known predisposition to medulloblastoma e.g. Gorlin's syndrome.

Ages: 4 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2004-04; Primary Completion 2008-12 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Free survival rate | 2 years after the start of the study
  To compare in a randomised trial the event free survival rate for children and adolescents with standard risk medulloblastoma treated with either hyperfractionated radiotherapy or reduced dose radiotherapy with conventional fractionation.

SECONDARY OUTCOMES:
To compare overall survival between the two treatment arms. | Follow-up of the last patient included up to the age of 20 years
  Will hyperfractionated radiotherapy lead to a different progression free (PFS) and overall survival (OS) compared to the standard arm radiotherapy?
To compare the pattern of relapse between the two treatment arms | Follow-up of the last patient included up to the age of 20 years
  Will hyperfractionated RT lead to a different pattern of local tumour control/pattern of relapse with particular respect to local relapse (tumour bed, posterior fossa outside the tumour bed) compared to the standard arm RT? The time to local progression should be the measure for the local tumour control.
To explore the benefit and the risks of neurosurgery | Follow-up of the last patient included up to the age of 20 years
  To determine the toxicity of surgery.To investigate whether there are identifiable factors that correlate with toxicity.
  To define the impact of any complications of surgery on commencement of adjuvant therapy and on EFS.

CONTACTS AND LOCATIONS:
Overall Officials: DOZ François, MD, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Derived] Goschzik T, Schwalbe EC, Hicks D, Smith A, Zur Muehlen A, Figarella-Branger D, Doz F, Rutkowski S, Lannering B, Pietsch T, Clifford SC. Prognostic effect of whole chromosomal aberration signatures in standard-risk, non-WNT/non-SHH medulloblastoma: a retrospective, molecular analysis of the HIT-SIOP PNET 4 trial. Lancet Oncol. 2018 Dec;19(12):1602-1616. doi: 10.1016/S1470-2045(18)30532-1. Epub 2018 Nov 1. PMID 30392813